CLINICAL TRIAL: NCT07162363
Title: Synergistic Intervention of Minimally Invasive Surgery and Deferoxamine in Intracerebral Hemorrhage (SMAD)
Brief Title: Synergistic Minimally Invasive Surgery and Deferoxamine in ICH
Acronym: SMAD
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY2025-0922
Record Dates: First submitted 2025-08-19; First posted 2025-09-09 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Intracerebral Hemorrhage; ICH - Intracerebral Hemorrhage
Keywords: deferoxamine; DFX; MIS; minimally invasive surgery; alteplase; ICH; Intracerebral hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Minimally Invasive Surgical Procedures; Deferoxamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MIS and IV Deferoxamine (Experimental): Patients in the investigational arm will receive intravenous deferoxamine (DFX) at 32 mg/kg per day, initiated within 1 hour of randomization and continued for 3 consecutive days. Once the hematoma is deemed stable for intervention, the MIS procedure will involve hematoma evacuation using different techniques tailored for superficial (lobar) and deep hemorrhages within 24 hours of Ictus.
  Interventions: Procedure: Minimally Invasive surgery (MIS); Drug: Deferoxamine
- Standard Medical Care (SMC) (Active Comparator): Participants will receive standard medical management for ICH without MIS or deferoxamine, serving as the control group.
  Interventions: Other: Standard Medical Care (SMD)

INTERVENTIONS:
Procedure: Minimally Invasive surgery (MIS) — Lobar (superficial) hematomas will be evacuated via a minimally invasive trans-sulcal parafascicular approach, whereas deep hematomas will be removed through a minimally invasive burr-hole approach with catheter placement to allow controlled clot dissolution using alteplase.
  Arms: MIS and IV Deferoxamine
Drug: Deferoxamine — Deferoxamine will be administered as a continuous intravenous infusion at a dose of 32 mg/kg/day over 24 hours for a total of 3 consecutive days.
  Other Names: Deferoxamine mesylate; Desferal
  Arms: MIS and IV Deferoxamine
Other: Standard Medical Care (SMD) — We will follow the American Heart Association and European Stroke Organization guidelines for the management of non-traumatic spontaneous intracerebral hemorrhage, ensuring a standardized approach to monitoring patients' airways, ventilation, intracranial pressure, sedation, and pharmacologic management of intracranial mass effect.
  Arms: Standard Medical Care (SMC)

SUMMARY:
This is a multicenter, randomized, open-label trial designed to evaluate the safety, feasibility, and efficacy of combining minimally invasive surgery (MIS) with intravenous deferoxamine (DFX) for the treatment of spontaneous intracerebral hemorrhage (ICH), compared to standard medical care.

This trial represents the first investigation of a dual-modality approach in ICH, integrating mechanical clot evacuation with biochemical neuroprotection, with the goal of improving neurological outcomes.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria:

1. Age ≥ 18 and ≤ 80 years
2. Spontaneous supratentorial ICH confirmed by CT or CTA, with hematoma volume:

   * ≥30 mL on initial diagnostic CT, OR
   * ≥25 mL on stability CT performed ≥6 hours after diagnostic CT,

     1. Clot growth must be less than 5 mL between scans to be eligible
     2. A second stability scan at least 12 hours later is allowed if clot expanded >5 mL
3. NIHSS score ≥ 6 at enrollment
4. Glasgow Coma Scale (GCS) score ≥5 and ≤14 at screening
5. Symptoms onset ≤ 24 hours before diagnostic CT

   * Use "last known well" for wake-up strokes
   * Unknown onset is exclusionary
6. SBP < 180 mm Hg sustained for at least 6 hours prior to randomization
7. Randomization must occur between 12 and 24 hours from initial diagnostic CT done at UIC or in case of transfers, at other institutions.
8. Functionally independent pre-ICH, defined as mRS 0-1. Pre-ICH functional status will be determined from medical records and structured interviews with the patient or a reliable caregiver, with ambiguous cases adjudicated by the site PI. Patients with mRS 0-1 are considered functionally independent, able to perform all usual activities without assistance.
9. Written informed consent obtained from patient or legal representative

Exclusion Criteria:

1. Infratentorial hemorrhage (e.g., brainstem or cerebellar hematoma).
2. Hemorrhage due to secondary causes: trauma, AVM, aneurysm, Moyamoya disease, hemorrhagic conversion of ischemic stroke, tumor, or vascular anomaly (diagnosed on imaging).
3. Recurrent ICH within the past year.
4. Intraventricular hemorrhage (IVH) requiring surgical treatment for trapped ventricle or mass effects (e.g., endoscopic evacuation). EVD is permitted.
5. Evidence of irreversible impaired brainstem function (e.g., bilateral fixed dilated pupils, decerebrate posturing).
6. Glasgow Coma Scale (GCS) ≤ 4 at screening, indicating extremely poor neurologic prognosis. NIHSS item 1a = 3, indicating comatose status (unresponsive to verbal or painful stimulation).
7. Thalamic ICH with midbrain extension and third nerve palsy.
8. Clinical indication for emergent surgical hematoma evacuation, as determined by treating neurosurgeons.
9. NIHSS score < 6 (too mild to benefit).
10. Expected withdrawal of care or death within 72 hours.
11. Prior enrollment in the study.
12. Creatinine ≥ 2.0 mg/dL or evidence of severe renal impairment.
13. Active hepatic failure or severe hepatic disease.
14. Pregnancy or breastfeeding.
15. Severe iron deficiency anemia (Hgb < 8 g/dL or ferritin <15 ng/mL).
16. Active systemic infection (e.g., sepsis, subacute bacterial endocarditis).
17. Active internal bleeding (GI, GU, retroperitoneal, pulmonary).
18. History of mechanical heart valve (bioprosthetic valves allowed).
19. Known left atrial/ventricular thrombus or high embolic risk (e.g., mitral stenosis + AFib).
20. Any coagulopathy:

    * Platelet count <100,000
    * INR > 1.4 not correctable within 6 hours
    * Use of NOACs (apixaban, rivaroxaban, dabigatran) or LMWH at presentation
21. Long-term anticoagulation that cannot be stopped safely (e.g., mechanical valve needing Coumadin).
22. Allergy or intolerance to DFX or rtPA.
23. Active alcohol or drug use that impairs adherence to follow-up.
24. Participation in another interventional trial. (Observational studies are allowed.
25. Inability or unwillingness to provide informed consent. This includes patients who lack decision-making capacity (and have no available legally authorized representative) or those who decline participation.
26. Not expected to survive to Day 365 or have DNR/DNI status at time of screening.
27. Any other condition that the investigator believes would pose a significant hazard or interfere with outcome assessments.
28. Patients with confirmed aspiration, pneumonia, pulmonary edema, evident bilateral pulmonary infiltrates on CXR or CT scan prior to enrollment.
29. Patients with significant respiratory disease such as chronic obstructive pulmonary disease, pulmonary fibrosis, or any use of chronic or intermittent inhaled O2 at home.
30. The presence of 4 or more of the following risk modifiers for ARDS prior to enrollment:

    1. Tachypnea (respiratory rate >30)
    2. SpO2 <95%
    3. Obesity, defined as Body Mass Index (BMI) >30 d) Acidosis (pH <7.35)

    e. Hypoalbuminemia (albumin <3.5 g/dL) f. Concurrent use of chemotherapy
31. Subjects who are taking prochlorperazine or are expected to undergo Gallium-67 imaging during the study period.
32. Known severe hearing loss.
33. Taking iron supplements containing ≥325 mg ferrous iron or prochlorperazine 34. Patients with heart failure taking >500 mg vitamin C daily

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Utility-weighted Modified Rankin Scale (mRS) | Post-randomization day 30, day 90, day 180
  The Modified Rankin Scale (mRS) is a standard measure of global disability after stroke or intracerebral hemorrhage. For this study, a utility-weighted mRS (uw-mRS) will be used to account for patient-centered quality-of-life differences across mRS levels. Higher utility scores indicate better functional outcomes. The uw-mRS will be assessed at Days 30, 90, and 180 after randomization to evaluate the long-term impact of the intervention on patient functional recovery.
Rate of All-Cause Mortality | Post-randomization day 30
  Percentage of participants who died from any cause within the first 30 days after randomization.
Rate of Procedure-Related Mortality | Post-randomization day 7
  Percentage of participants who died due to the study procedures within the first 7 days after randomization.
Rate of Infectious Complications | Post-randomization day 30
  Percentage of participants who developed a bacterial brain infection (cerebritis, meningitis, or ventriculitis) within 30 days of randomization.
Other Adverse Events | Post-randomization day 30
  Percentage of participants experiencing adverse events related to allergic reactions, cardiovascular events (hypotension, tachycardia), renal or hepatic dysfunction, or seizures.
Rate of Procedural Complications | Post-randomization day 30
  Percentage of participants with cerebrospinal fluid (CSF) leaks or other surgery-related complications requiring intervention.
Rate of Symptomatic Intracranial Hemorrhage | Post-randomization day 7
  Percentage of participants experiencing symptomatic rebleeding or hematoma expansion within 7 days of post-randomization.

SECONDARY OUTCOMES:
Hematoma and Edema Volume on Imaging | From randomization until end of treatment (up to 10 days) for early response, and at 30-, 90-, and 180-days post-randomization for follow-up assessments.
  Early Treatment Response: Percentage of hematoma resolved at the end-of-treatment CT scan compared with the stability CT scan performed prior to randomization.
  Follow-Up Assessment: Percentage of hematoma and perihematomal edema resolved on CT scans performed at 30, 90, and 180 days compared with both the stability CT scan and the end-of-treatment CT scan.
Intensive Care Unit (ICU) and Hospital Length of Stay | Within 3 months after randomization
  Total length of initial ICU and hospital stay within 3 months after randomization
Mortality | Post-treatment day 180

CONTACTS AND LOCATIONS:
Overall Officials: Gursant S. Atwal, MD, Principal Investigator — University of Illinois Hospital & Health Sciences System (UI Health); Javed Iqbal, MBBS, Study Director — University of Illinois Hospital & Health Sciences System (UI Health)
Locations (1):
- University of Illinois Hospital & Health Sciences System (UI Health), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided